CLINICAL TRIAL: NCT07375602
Title: Multimodal Clinical Data Integration and Artificial Intelligence Modeling for Predicting Complications Following Pediatric Transcatheter Closure of Perimembranous Ventricular Septal Defect
Brief Title: A Multimodal AI Prediction Model for Complications After Transcatheter Closure of Perimembranous VSD in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kun Sun, Professor of Department of Pediatric Cardiology, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XHEC-C-2025-295-1
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Disease (CHD); Ventricular Septal Defects (VSD); Cardiac Catheterization; Postoperative Complications
MeSH Terms: conditions — Heart Defects, Congenital; Heart Septal Defects, Ventricular; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to develop and validate a multimodal artificial intelligence prediction model for treatment-related complications in children with perimembranous ventricular septal defect (pmVSD) undergoing transcatheter device closure. The main question it aims to answer is: Can an AI model that integrates demographics, laboratory results, electronic health record text, echocardiography reports, chest radiographs, and electrocardiogram accurately predict the risk of complications at the individual patient level? Data will be retrospectively collected from routine clinical care records of pediatric patients who underwent transcatheter closure for pmVSD. Deep learning methods will be used to extract features from text and images to train and validate the prediction model.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 18 years at the time of transcatheter procedure.
* Diagnosis of perimembranous ventricular septal defect confirmed by echocardiography, and underwent transcatheter device closure at the study center.
* Medical records sufficient to ascertain the primary outcome within the pre-specified follow-up window, and availability of minimum baseline clinical information required for model development/validation.

Exclusion Criteria:

* Ventricular septal defects not classified as perimembranous on echocardiography, including muscular, outlet, or inlet VSDs, as well as multiple or complex VSDs involving more than one septal region.
* Presence of complex congenital heart disease or associated structural abnormalities requiring concomitant surgical repair (e.g., tetralogy of Fallot).
* Prior surgical VSD repair or prior transcatheter VSD closure.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (18 years or younger) with echocardiography-confirmed perimembranous ventricular septal defect who underwent transcatheter device closure at Xinhua Hospital between January 1, 2015, and December 31, 2025, identified retrospectively from routine clinical care records.
Sampling Method: Probability Sample
Enrollment: 5249 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Composite Procedure-Related Complications After Transcatheter Closure of Perimembranous VSD | Up to 30 Days After Transcatheter Closure
  Occurrence of a composite endpoint of procedure-related complications, including arrhythmia requiring treatment, new-onset or worsened valvular regurgitation, residual shunt requiring reintervention, and device embolization.

SECONDARY OUTCOMES:
Area Under the Precision-Recall Curve (AUCPR) for Complication Prediction | Up to 30 Days After Transcatheter Closure
  The area under the precision-recall curve (AUCPR) of the model for predicting the primary composite procedure-related complication endpoint.
Sensitivity of the Model at a Pre-Specified Risk Threshold | Up to 30 Days After Transcatheter Closure
  Sensitivity for predicting the primary composite procedure-related complication endpoint at a pre-specified probability (risk) threshold.
Positive Predictive Value (PPV) of the Model at a Pre-Specified Risk Threshold | Up to 30 Days After Transcatheter Closure
  Positive predictive value (PPV) for predicting the primary composite procedure-related complication endpoint at the same pre-specified probability (risk) threshold.
Negative Predictive Value (NPV) of the Model at a Pre-Specified Risk Threshold | Up to 30 Days After Transcatheter Closure
  Negative predictive value (NPV) for predicting the primary composite procedure-related complication endpoint at the same pre-specified probability (risk) threshold.

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be made publicly available due to privacy considerations and institutional data governance policies for retrospective electronic health record and imaging data. Aggregated results may be shared in publications and presentations.